CLINICAL TRIAL: NCT03513718
Title: Incidence of Acute Kidney Injury After Cardiac Surgery on Cardiopulmonary Bypass in the Pediatric Intensive Care Unit of Lausanne. A Retrospective Study
Brief Title: Acute Kidney Injury After Cardiac Surgery on CPB
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Perez Maria-Helena, MD, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 2017-01542
Record Dates: First submitted 2018-04-09; First posted 2018-05-01 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Acute Kidney Injury; Congenital Heart Disease; Surgery; CBP; Child, Only
Keywords: Acute kidney injury, AKI
MeSH Terms: conditions — Acute Kidney Injury; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this retrospective study is to determine the incidence and severity of acute kidney injuries (AKI) after heart surgery on cardiopulmonary bypass (CPB) in the pediatric intensive care unit (PICU) in Lausanne, Switzerland.

DETAILED DESCRIPTION:
The investigators will review in a retrospective way, all patients aged between 0 and 16 years, admitted in the PICU after cardiac surgery on CPB from 01.01.2014 to 31.12.2016. They will asses for AKI. The first step is to determine the incidence and severity, the second step is to determine the risk factors for AKI and/or protecting factors.

ELIGIBILITY:
Inclusion Criteria:

- all pediatric patients (0-16 years) admitted to PICU after cardiac surgery with CPB.

Exclusion Criteria:

* Preexisting kidney injury,
* no preoperative creatinine lab value

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Retrospective inclusion of all pediatric patients (0-16 years) admitted in our PICU after cardiac surgery with CPB between January 2014 and December 2016
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Presence and severity of an AKI occurring during stay in the PICU | up to 3 month
  Scoring AKI with pRiffle

SECONDARY OUTCOMES:
PICU stay and ventilation time | up to 3 month
  correlation between AKI and invasive ventilation/duration and PICU stay
Persisting AKI after release from PICU according to RIFLE score | more than 3 month
  After leaving ICU

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Hélène Perez, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
No sharing of patients data